CLINICAL TRIAL: NCT05891093
Title: A Prospective, Randomized, Open-label Phase III Clinical Study of the Efficacy and Safety of Fluzoparib Combined With Adjuvant Endocrine Therapy Versus Adjuvant Endocrine Therapy for HR+/HER2- SNF3-subtype Early Breast Cancer (BCTOP-L-A01)
Brief Title: Efficacy and Safety of Fluzoparib Combined With Adjuvant Endocrine Therapy for HR+/HER2- SNF3-subtype Early Breast Cancer (BCTOP-L-A01)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Chief Physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N056
Record Dates: First submitted 2023-05-24; First posted 2023-06-06 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: fluzoparib; adjuvant treatment; SNF3-subtype
MeSH Terms: conditions — Breast Neoplasms | interventions — fluzoparib; Anastrozole; Letrozole; exemestane; Tamoxifen; Toremifene; abemaciclib; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluzoparib+Endocrine Therapy (Experimental): Fluzoparib 50mg bid orally for 1 year, combined with physician's choice of endocrine therapy as clinically indicated (eg, aromatase inhibitor, tamoxifen, toremifene endocrine therapy for 5 to 10 years; CDK4/6 inhibitor therapy for 2 years; ovarian function suppression with LHRH agonist).
  Interventions: Drug: Fluzoparib; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Tamoxifen; Drug: Toremifene; Drug: Abemaciclib; Drug: LHRH agonist
- Endocrine Therapy (Active Comparator): Physician's choice of endocrine therapy as clinically indicated (eg, aromatase inhibitor, tamoxifen, toremifene endocrine therapy for 5 to 10 years; CDK4/6 inhibitor therapy for 2 years; ovarian function suppression with LHRH agonist).
  Interventions: Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Tamoxifen; Drug: Toremifene; Drug: Abemaciclib; Drug: LHRH agonist

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib 50mg bid orally for 1 year.
  Arms: Fluzoparib+Endocrine Therapy
Drug: Anastrozole — 1mg, qd orally
Drug: Letrozole — 2.5mg, qd orally
Drug: Exemestane — 25mg, qd orally
Drug: Tamoxifen — 10mg, bid orally
Drug: Toremifene — 60mg, qd orally
Drug: Abemaciclib — 150mg/100mg/50mg, bid orally for 2 years
Drug: LHRH agonist — Leuprorelin acetate, goserelin acetate

SUMMARY:
This is a prospective, randomized, open-label phase III clinical study on the efficacy and safety of fluzoparib combined with adjuvant endocrine therapy versus adjuvant endocrine therapy for HR+/HER2- SNF3-subtype early breast cancer.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label phase III clinical study on the efficacy and safety of fluzoparib combined with adjuvant endocrine therapy versus adjuvant endocrine therapy for HR+/HER2- SNF3-subtype early breast cancer.

A total of 766 patients with luminal-type early breast cancer who received surgery at the Fudan University Shanghai Cancer Cancer and were classified as SNF3 (proliferative) by SNF algorithm fusion clustering will be collected for this study. Before enrollment, the primary tumors of the patients were subjected to molecular typing based on H&E slices combined with digital pathology, and subsequent enrollment could be considered if patient pathology was confirmed as SNF3 subtype.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-70 years old;
2. ECOG score 0 or 1;
3. ER+/HER2- confirmed by histopathology after early breast cancer surgery（ER positive is defined as immunohistochemistry(IHC) detection of ER ≥ 1% HER2-negative is defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (Fluorescence in situ hybridization (FISH), Chromogenic in situ hybridization (CISH) , or Silver in situ hybridization (SISH)) test is required by local laboratory testing.); definition of SNF3 subtype: SNF3 subtype confirmed by digital pathology of H&E sections;
4. Postoperative pathological stage T2-4N0-3M0;
5. Patients who have previously received neoadjuvant chemotherapy and/or adjuvant chemotherapy;
6. Time of randomization from surgery does not exceed 16 months;
7. Time of endocrine therapy from last non-endocrine anti-tumor treatment does not exceed 12 weeks;
8. Has adequate organ function meeting the following criteria: (1) adequate bone marrow function: hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); absolute neutrophil count ≥ 1.5 x 10^9 /L; platelet count ≥ 100 * 10^9 /L; (2)adequate liver and kidney function: Alanine Aminotransferase (ALT) ≤ 3×upper limit of normal (ULN), Aspartate Aminotransferase (AST) ≤ 3×ULN, Total Bilirubin (TBIL)≤ 1.5×ULN, serum creatinine ≤ 1×ULN，and with endogenous creatinine clearance rate of >50 ml/min (Cockcroft-Gault formula);
9. Patients receiving radiotherapy must recover from the acute phase reaction of radiotherapy, with a washout period of at least 14 days from the end of radiotherapy to randomization;
10. Patients who received chemotherapy in the early stage must recover from acute adverse reactions to chemotherapy ([CTCAE] grade ≤ 1) before randomization, except for hair loss or grade 2 peripheral neuropathy. There is a washout period of at least 21 days from the last chemotherapy administration to randomization (assuming the patient has not received radiotherapy);
11. Patients can take medication orally on their own;
12. Female subjects with fertility are required to use a medically approved contraceptive method during the study treatment
13. Participants voluntarily joined the study, has signed informed consent before any trial related activities are conducted, has good compliance and has agreed to follow-up.

Exclusion Criteria:

1. Has bilateral breast cancer;
2. Has previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ.
3. Has metastatic (Stage 4) breast cancer;
4. Is pregnant, is breast feeding women, or women of childbearing age who cannot practice effective contraceptives;
5. Patients participating in other clinical trials at the same time;
6. Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous of randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmgh, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension;
7. Has known allergy to fluzoparib and excipients.
8. Has severe or uncontrolled infection;
9. Has a history of psychotropic substance abuse and were unable to abandon drug habits, or those with history of mental disorders;
10. The researchers judged patients to be unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
invasive disease free survival (iDFS) | 5 years
  defined as occurrence of any of the following: ipsilateral invasive breast cancer recurrence, regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer, or second non-breast invasive cancer.In-situ events are not included.

SECONDARY OUTCOMES:
distant relapse free survival (DRFS) | 5 years
  the time from operation to the first distant recurrence, and the cases of death without distant recurrence was censored at the time of the death
overall survival (OS) | 5 years
  the time from treatment to death, regardless of disease recurrence
Adverse Effects | 5 years
  an undesired harmful effect resulting from a medication or other intervention
Number of participants with Patient Reported Outcome (PRO) | 5 years
  a health outcome directly reported by the patient who experienced it.

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Academy of Medical Sciences Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangdong, Guangzhou
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang